CLINICAL TRIAL: NCT03889171
Title: Predisposition to Breast Cancer BRCA1 / BRCA2 and to HNPCC Colon : Comparison to Psychological, Medical and Emotional Influencing Communication and Achievement Factors to Oncogenetics Tests
Brief Title: Comparison to Psychological, Medical and Emotional Influencing Communication and Achievement Factors to Oncogenetics Tests
Acronym: PSICOM
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8893
Record Dates: First submitted 2019-03-11; First posted 2019-03-26 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Cancer; Colorectal Cancer; Breast Cancer; Ovarian Cancer
Keywords: genetic testing; genes BRCA1; genes BRCA2; mutation; family; disclosure; psychology; DNA mismatch repair; genetic predisposition to disease; cancer; oncology
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Fanconi Anemia, Complementation Group D1; Genetic Predisposition to Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Behaviour — Comparison to psychological, medical and emotional Influencing communication and achievement factors to Oncogenetics tests

SUMMARY:
The purpose of the study was to analyze the psychological and emotional determinants of domestic dissemination of information about genetic risk of cancer and to compare the level of diffusion syndromes in breast/ ovarian cancer ( BRCA1 / BRCA2) and colon/endometrial ( HNPCC )

DETAILED DESCRIPTION:
The risk associated with a genetic predisposition is among the various forms of risk, the strongest identifiable risk . It enables to offer people at risk an appropriate medical care (screening, prevention ) the clinical benefit is validated today. The person with whom a predisposing mutation has been identified must communicated its related information on the risk of cancer and the ability to perform genetic analysis. It appears that this dissemination of information is not always optimal, as shown in figures from the National Cancer Institute joined the project; the purpose of the study was to analyze the psychological and emotional determinants of domestic dissemination of information about genetic risk of cancer and to compare the level of diffusion syndromes in breast/ ovarian cancer ( BRCA1 / BRCA2) and colon/endometrial ( HNPCC )

ELIGIBILITY:
Inclusion Criteria:

* Patient having a deleterious genetic mutation on genes BRCA1 and/or BRCA2 and or on genes MMR
* The patient being of the family (who carried out a full analysis of BRCA1/BRCA2 and/or those MMR )

Exclusion Criteria:

* Patient not carrying a deleterious genetic mutation on the BRCA1/2 genes and/or those of the MMR system,
* Patient under guardianship, curator or unable to give his non-opposition,
* Adult patients protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female and male participants are being studied
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
intrafamilial disclosure rate | On average 1 year
  The intrafamilial disclosure rate assessed the number of relatives informed by the proband about the mutation (according to the proband) out of the number of relatives at risk of carrying the familial mutation. Relatives who were considered "at risk" were first, second, third or fourth-degree relatives, older than 18 years and related to the relevant side of the family or, if unknown, just related to the proband whatever the family side.
relatives' genetic targeted testing uptake rate | On average 1 year
  The relatives' genetic targeted testing uptake rate assessed the number of relatives considered by the proband to have taken up the genetic targeted testing out of the number of relatives informed by the proband. To assess the potential bias of the proband's perception of genetic targeted testing uptake by relatives, we compared the number of relatives who underwent genetic targeted testing according to the proband with the number of tests actually performed. This anonymous comparison was performed in a subset of the population within the geographic regional area of Montpellier where all analyses are centralized in a single laboratory. Probands were asked how many relatives living in the region underwent genetic testing and this number was compared with the information available from the University Laboratory of Montpellier.

IPD SHARING:
Plan to Share IPD: Undecided